CLINICAL TRIAL: NCT00571987
Title: Pilot Study of Radiofrequency Ablation of Breast Cancer Lumpectomy Sites to Decrease Re-operation
Acronym: eRFA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAMS 29143
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Results first posted 2015-10-06 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-10

CONDITIONS: Cancer of the Breast
Keywords: Breast cancer; Lumpectomy; Radiofrequency Ablation; Negative margins; Breast Conserving Surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): This is a non-randomized one arm study, all subjects receive treatment (radiofrequency ablation).
  Interventions: Device: AngioDynamics (previously RITA Med,Inc) radiofrequency delivery system (consisting of a generator and Starburst XL probe)

INTERVENTIONS:
Device: AngioDynamics (previously RITA Med,Inc) radiofrequency delivery system (consisting of a generator and Starburst XL probe) — Generator is connected to a single use probe. Probe is inserted into the lumpectomy cavity and heated to 100 degrees Celsius and held there for 15 minutes, after which probe is removed.

SUMMARY:
In this protocol we combine two available and reliable treatments - lumpectomy and RFA. This combination method will provide for excision of the cancer as routinely accomplished and ablation of the cancer bed (lumpectomy site) to ensure negative margins without removing large volumes of tissue. This combined open technique will allow for full histologic analysis of the primary tumor and margin. Because no extra tissue is removed from the breast to generate negative margins it will result in better cosmesis than re-excision to obtain negative margins.

DETAILED DESCRIPTION:
While RFA alone is not approved for tumor destruction in breast it is FDA-approved for ablation of soft tissue after the breast cancer is removed. This study seeks to remove the tumor and then ablate a tumor-free zone (margin) of tissue around the lumpectomy site instead of removing more tissue. The primary short-term goal is to obviate the need for re-excision in the event of close or positive margins (< 3 mm) which occurs on average in ~40 percent of the cases. Permanent pathology is only an estimation of margin status since 90% of recurrences occur at the site of the original lumpectomy. RFA ensures a sterilized margin regardless of the accuracy of the permanent pathology.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18-100 years old
* Not pregnant or breastfeeding
* Pre-study radiologic documentation of:
* size ≤ 5 cm
* unicentric, unilateral
* suspicious mass or calcification
* BIRADS classification ≥ IV
* location of abnormality > 1 cm from skin
* Ductal or Infiltrating Ductal Carcinoma
* Grade I-III on final pathology
* Good general health
* Zubrod Performance Status of 0,1, or 2
* No previous chemotherapy
* No palpable axillary or supraclavicular lymph nodes
* If prior non-breast malignancy, must have > 5 year disease-free survival

Exclusion Criteria:

* Patient < 18 y/o or > 100 y/o
* Pregnant or breastfeeding
* Male
* Breast implants
* Multicentric disease or bilateral disease
* Lesions > 5 cm in diameter
* Lesions < 1.0 cm from the skin
* Previous prior radiation to the breast
* Need for mastectomy
* Diffuse microcalcifications (as determined by the Investigator)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2004-09; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: V. Suzanne Klimberg, M.D., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas For Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Background] Klimberg VS, Kepple J, Shafirstein G, Adkins L, Henry-Tillman R, Youssef E, Brito J, Talley L, Korourian S. eRFA: excision followed by RFA-a new technique to improve local control in breast cancer. Ann Surg Oncol. 2006 Nov;13(11):1422-33. doi: 10.1245/s10434-006-9151-4. Epub 2006 Sep 29. PMID 17009144
- [Background] Klimberg VS, Boneti C, Adkins LL, Smith M, Siegel E, Zharov V, Ferguson S, Henry-Tillman R, Badgwell B, Korourian S. Feasibility of percutaneous excision followed by ablation for local control in breast cancer. Ann Surg Oncol. 2011 Oct;18(11):3079-87. doi: 10.1245/s10434-011-2002-y. Epub 2011 Sep 9. PMID 21904959
- [Background] Mackey A, Feldman S, Vaz A, Durrant L, Seaton C, Klimberg VS. Radiofrequency ablation after breast lumpectomy added to extend intraoperative margins in the treatment of breast cancer (ABLATE): a single-institution experience. Ann Surg Oncol. 2012 Aug;19(8):2618-9. doi: 10.1245/s10434-012-2293-7. Epub 2012 Mar 16. PMID 22422482
- [Background] Klimberg VS, Ochoa D, Henry-Tillman R, Hardee M, Boneti C, Adkins LL, McCarthy M, Tummel E, Lee J, Malak S, Makhoul I, Korourian S. Long-term results of phase II ablation after breast lumpectomy added to extend intraoperative margins (ABLATE l) trial. J Am Coll Surg. 2014 Apr;218(4):741-9. doi: 10.1016/j.jamcollsurg.2013.12.032. Epub 2014 Jan 11. PMID 24655863
- See also: Long-Term Results of Phase II Ablation after Breast Lumpectomy Added to Extend Intraoperative Margins (ABLATE l) Trial Presented at the Southern Surgical Association 125th Annual Meeting, Hot Springs, VA, December 2013. — http://dx.doi.org/10.1016/j.jamcollsurg.2013.12.032

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was consented to the study in September 2004. The final subject was consented in March 2010. A total of 107 subjects were consented.
Pre-assignment Details: As part of this non-blinded and non-randomized study all participants receive ablation.
Groups:
- Subjects Received RFA Treatment: AngioDynamics (previously RITA Med,Inc) radiofrequency delivery system (consisting of a generator and Starburst XL probe): Generator is connected to a single use probe. Probe is inserted into the lumpectomy cavity and heated to 100 degrees Celsius and held there for 15 minutes, after which probe is removed.
Period: Overall Study
Arm/Group | Subjects Received RFA Treatment
Started | 107
Completed | 100
Not Completed | 7

BASELINE CHARACTERISTICS:
Groups:
- RFA Treatment: AngioDynamics (previously RITA Med,Inc) radiofrequency delivery system (consisting of a generator and Starburst XL probe): Generator is connected to a single use probe. Probe is inserted into the lumpectomy cavity and heated to 100 degrees Celsius and held there for 15 minutes, after which probe is removed.
Arm/Group | RFA Treatment
Number analyzed (Participants) | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.02 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Requiring 2nd Surgery for Close or Positive Margins
Description: A "close" surgical margin implies that cancer cells are found on pathology to be very close to the surgical margin, and a "wide" surgical margin implies the tumor exists far from the cut edge or the surgical margin. For this study, we defined "close" as less than 3 mm.
Time Frame: Margins assessed at Final Pathology, approximately 1 week post-RF surgery
Measure: Number; unit: participants
Groups:
- Margin Status: AngioDynamics (previously RITA Med,Inc) radiofrequency delivery system (consisting of a generator and Starburst XL probe): Generator is connected to a single use probe. Probe is inserted into the lumpectomy cavity and heated to 100 degrees Celsius and held there for 15 minutes, after which probe is removed.
Arm/Group | Margin Status
Number analyzed (Participants) | 100
participants | 22

2. Secondary Outcome: Recurrence of Breast Cancer at Prior Site of Disease
Time Frame: Until study end (2 years)
Population: During the 68-month median follow-up in patients not treated with XRT, there were 2 in-site tumor recurrences treated with AI, 3 biopsy entrance site recurrences treated with excision and XRT to conserve the breast, and 2 recurrences elsewhere and 1 contralateral recurrence; all 3 treated with mastectomy.
Measure: Number; unit: participants
Groups:
- Recurrences at the Site: AngioDynamics (previously RITA Med,Inc) radiofrequency delivery system (consisting of a generator and Starburst XL probe): Generator is connected to a single use probe. Probe is inserted into the lumpectomy cavity and heated to 100 degrees Celsius and held there for 15 minutes, after which probe is removed.
Arm/Group | Recurrences at the Site
Number analyzed (Participants) | 100
participants | 2

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | RFA Treatment
Serious Adverse Events (participants affected / at risk) | 0/107
Other Adverse Events (participants affected / at risk) | 9/107
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RFA Treatment (N=107)
Wound complication (Skin and subcutaneous tissue disorders) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No